CLINICAL TRIAL: NCT02414087
Title: Therapeutic Effects of Customized Insoles on Children With Flat Foot
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Shin Kong Wu Ho-Su Memorial Hospital, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SKH-8302-104-DR-29
Record Dates: First submitted 2015-03-27; First posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Flat Foot
Keywords: flat foot; therapeutic effect; insoles; children
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Active Comparator): ICB Medical Insoles
  Interventions: Device: ICB Medical insoles
- control group (Placebo Comparator): without ICB Medical insoles

INTERVENTIONS:
Device: ICB Medical insoles — Study group:
  Participants in the study group will be prescribed with customized full-length insoles (ICB Medical) to keep the subtalar joint in neutral position, using self chosen comfortable shoes, for 3 months.
  Control group:
  Participants in the control group will not be prescribed with customized full-length insoles (ICB Medical) to keep the subtalar joint in neutral position, using self chosen comfortable shoes, for 3 months
  Arms: study group

SUMMARY:
Using double blind, randomized controlled design to study the short-term therapeutic effects of customized arch-support shoe insoles to children with flat foot.

DETAILED DESCRIPTION:
A total of 52 children with flat foot will be collected. The participants will be randomized into two groups, including study group (insoles group) and control group (without insole group).

All participants in the insoles group will be evaluated at baseline, that is before the customized full-length shoe insoles are prescribed. All the evaluations, including physical functional ability, balance, physical activity, functional performance, and quality of life will be re-evaluated up to 12 weeks after shoe insoles wearing in the insoles group.

The control group will be evaluated at the baseline and up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* flat foot

Exclusion Criteria:

* age less than 3 years old or older than 10 years old
* pathological flat foot

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
health related quality of life (Pediatric Quality of Life Inventory (PedQoL) | baseline and up to 12 weeks
  Pediatric Quality of Life Inventory (PedQoL)

SECONDARY OUTCOMES:
functional performance (Pediatric Outcome Data Collection Instrument) | baseline and up to 12 weeks
  Pediatric Outcome Data Collection Instrument

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital; Taipei Medical University
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 26;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub4. PMID 35080267
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 14;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub3. PMID 35029841